CLINICAL TRIAL: NCT02498925
Title: Examining Reward-Related Predictors and Mechanisms of Change in BA Treatment for Anhedonic Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christian A. Webb, Associate Professor, Harvard Medical School; Associate Psychologist, McLean Hospital, Mclean Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-D000149; K23MH108752 (NIH)
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anhedonic teens receiving Behavioral Activation (BA) (Experimental): 12 weeks (1 50-min session per week) of Behavioral Activation for the anhedonic adolescents.
  Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral strategies to improve mood and places little emphasis on cognitive restructuring techniques.
  Interventions: Behavioral: Behavioral Activation
- Non-anhedonic teens (not receiving BA) (No Intervention): A group of adolescents with no anhedonia were recruited

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral change strategies to improve mood and places little emphasis on cognitive restructuring techniques.
  Arms: Anhedonic teens receiving Behavioral Activation (BA)

SUMMARY:
The prevalence of major depressive disorder (MDD) is relatively low in childhood (i.e., 1-3%), but increases substantially during adolescence. By the age of 18, approximately 15% of adolescents will have experienced at least one episode of MDD. A growing body of research implicates abnormalities in reward circuitry as playing a critical role in the development and maintenance of depressive symptoms in adolescents. Importantly, these reward-circuitry abnormalities have been linked to anhedonia (i.e., decreased pleasure or blunted reactivity to rewarding stimuli). Behavioral Activation (BA) represents a promising - and relatively simple to deliver - nonpharmacologic intervention for adolescent depression, which has been shown to be at least as effective as Cognitive Behavioral Therapy (CBT) with regards to symptom reduction and lowering the risk of relapse in adult samples. More recently, promising data have emerged from the application of BA to depressed adolescents. BA can be conceptualized as a treatment directly targeting anhedonia. More specifically, BA targets anhedonia through behavioral change strategies aimed at gradually increasing patients' exposure to and engagement with rewarding stimuli and positively reinforcing experiences. Given this treatment focus, BA may be particularly beneficial for adolescents struggling with relatively elevated levels of anhedonic symptoms. Accordingly, the present study will examine the role of anhedonia and reward functioning in predicting treatment response in BA. In addition, analyses will be conducted examining the reward-related neural and behavioral mechanisms underlying anhedonic symptom improvement in BA.

DETAILED DESCRIPTION:
Participants in this research will include 35 anhedonic adolescents and 35 demographically matched healthy participants recruited from the greater Boston community by Dr. Webb at McLean Hospital's Center for Depression, Anxiety and Stress Research. The anhedonic adolescents will undergo 12 weeks of Behavioral Activation therapy. This study will include three sessions:

* The first session will involve a diagnostic interview, and a series of questionnaires and assessments.
* The second session will take place at the McLean Hospital's Neuroimaging Center, and involve an fMRI brain scan and administration of two behavioral tasks, as well as questionnaires.
* Following the 12-weeks treatment, anhedonic adolescents will return to McLean Hospital's Neuroimaging Center for an fMRI brain scan, two behavioral tasks, and questionnaires. The healthy control group will complete the same three assessments at corresponding time points.

ELIGIBILITY:
General Inclusion Criteria:

* Both genders, any ethnicity
* Ages 13-18
* English as first language or English fluency
* Right handed
* Smartphone with iOS or Android platform (for EMA)
* Anhedonic Sample: Total Snaith Hamilton Pleasure Scale (SHAPS) score ≥ 3; Healthy Control Sample: Total SHAPS score = 0

General Exclusion Criteria:

* History of head trauma with loss of consciousness
* History of seizure disorder
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of cocaine or stimulant use (e.g., amphetamine, cocaine, methamphetamine)
* History of use of dopaminergic drugs (including methylphenidate)
* Clinical or laboratory evidence of hypothyroidism
* Systemic medical or neurological illness that could impact fMRI measures of cerebral blood flow
* Meet standard exclusion criteria for fMRI scanning (e.g. claustrophobia, cardiac pacemakers, neural pacemakers, surgically implanted metal devices, cochlear implants, metal braces, or other metal objects in their body);
* Positive urine pregnancy test

A. Anhedonic Adolescents:

Additional Exclusion Criteria:

* Subjects with suicidal ideation where outpatient BA treatment is determined unsafe or inappropriate by the study clinician. These patients will be immediately referred to appropriate clinical treatment
* History or current diagnosis of any of the following DSM-5 psychiatric illnesses: schizophrenia spectrum or other psychotic disorder, bipolar disorder, OCD, PTSD, substance (including alcohol) use disorder within the past 12 months or lifetime severe substance use disorder (i.e., meeting former DSM-IV criteria for past substance dependence). Simple phobia, social anxiety disorder, panic disorder, and generalized anxiety disorder will be allowed only if secondary to anhedonia
* Meet criteria for chronic depression (current episode > 2 years)
* Currently receiving psychotropic treatment or psychotherapy
* Absence of any psychotropic medications: 8 weeks for fluoxetine, 4 weeks for neuroleptics, 8 weeks for benzodiazepines, 6 weeks any other antidepressants

B. Healthy Control Adolescents:

Additional Exclusion Criteria:

* Elevated depressive symptoms as assessed in phone screen
* History of meeting criteria for any DSM-5 psychiatric or substance-related disorder
* Use of any psychiatric medications
* Family history (first-degree relatives) of any psychiatric disorder

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2022-04 (Actual); Study Completion 2023-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Webb, Ph.D., Principal Investigator — McLean Hospital & McLean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Result] Webb CA, Murray L, Tierney AO, Forbes EE, Pizzagalli DA. Reward-related predictors of symptom change in behavioral activation therapy for anhedonic adolescents: a multimodal approach. Neuropsychopharmacology. 2023 Mar;48(4):623-632. doi: 10.1038/s41386-022-01481-4. Epub 2022 Oct 28. PMID 36307561
- [Result] Webb CA, Murray L, Tierney AO, Gates KM. Dynamic processes in behavioral activation therapy for anhedonic adolescents: Modeling common and patient-specific relations. J Consult Clin Psychol. 2024 Aug;92(8):454-465. doi: 10.1037/ccp0000830. Epub 2023 Jun 5. PMID 37276084
- [Result] Ren B, Balkind EG, Pastro B, Israel ES, Pizzagalli DA, Rahimi-Eichi H, Baker JT, Webb CA. Predicting states of elevated negative affect in adolescents from smartphone sensors: a novel personalized machine learning approach. Psychol Med. 2023 Aug;53(11):5146-5154. doi: 10.1017/S0033291722002161. Epub 2022 Jul 27. PMID 35894246
- [Derived] Fisher H, Jaffe NM, Rahimi-Eichi H, Forbes EE, Pizzagalli DA, Baker JT, Webb CA. Measuring activation during behavioral activation therapy: a proof-of-concept study using smartphone sensors and LLM-derived ratings in adolescents with anhedonia. NPP Digit Psychiatry Neurosci. 2025 Oct 13;3:24. doi: 10.1038/s44277-025-00045-w. eCollection 2025. PMID 41098338

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Activation: 12 weeks (1 50-min session per week) of Behavioral Activation for the anhedonic adolescents.
  Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral strategies to improve mood and places little emphasis on cognitive restructuring techniques.
  Behavioral Activation: Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral change strategies to improve mood and places little emphasis on cognitive restructuring techniques.
- Non-anhedonic Adolescents: Non-anhedonic (healthy control) adolescents who did not receive behavioral activation (BA)
Period: Overall Study
Arm/Group | Behavioral Activation | Non-anhedonic Adolescents
Started | 39 | 41
Completed | 34 | 35
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Population: 39 anhedonic and 41 non-anhedonic
Groups:
- Anhedonic Adolescents Receiving Behavioral Activation: 12 weeks (1 50-min session per week) of Behavioral Activation for the anhedonic adolescents.
  Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral strategies to improve mood and places little emphasis on cognitive restructuring techniques.
  Behavioral Activation: Behavioral Activation is a psychosocial treatment for depression focused on gradually re-engaging patients with sources of reinforcement and reward in their environment (e.g., increasing activites and interpersonal interactions). In contrast to Cognitive Behavioral Therapy, and as the name implies, Behavioral Activation focuses on behavioral change strategies to improve mood and places little emphasis on cognitive restructuring techniques.
- Non-Anhedonic Adolescents: Adolescents without anhedonia (healthy controls) who did not receive behavioral activation
- Total: Total of all reporting groups
Arm/Group | Anhedonic Adolescents Receiving Behavioral Activation | Non-Anhedonic Adolescents | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.7 (1.9) | 16.2 (1.7) | 15.9 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 55
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 6 | 7
  White | 32 | 29 | 61
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80
Snaith-Hamilton Pleasure Scale (SHAPS) [Mean (Standard Deviation); unit: SHAPS total score] — A measure of anhedonia
  SHAPS total score | 36.18 (5.85) | 17.85 (3.91) | 26.79 (10.45)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anhedonic (Snaith-Hamilton Pleasure Scale; SHAPS) Symptoms
Description: Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item questionnaire that measures the capacity to experience pleasure (lack of pleasure is referred to as anhedonia). Total scores range from 14-56 with higher scores reflecting more anhedonia
Time Frame: Change from pre-treatment (baseline) to post-treatment (12 weeks)
Population: Participants who completed pre- and post-treatment SHAPS (and corresponding timepoints for non-anhedonic control group who did not receive BA treatment)
Measure: Mean (Standard Deviation); unit: units on SHAPS scale
Groups:
- Non-anhedonic Adolescent Control Group: Non-anhedonic (healthy control) adolescents who did not receive behavioral activation
Arm/Group | Behavioral Activation | Non-anhedonic Adolescent Control Group
Number analyzed (Participants) | 34 | 35
units on SHAPS scale | 7.06 (8.65) | -1.29 (3.57)

2. Primary Outcome: Change in Brain (Striatal and Medial PFC) Activation During a Monetary Reward Gambling Task
Description: During the pre- and post-treatment fMRI scan, youth completed an event-related card- guessing task designed to assess brain responses to the anticipation and receipt of monetary reward and loss. The task included four 6.5-min blocks in which youth guessed whether the value of a card was higher or lower than 5. Based on the trial type (win, loss, neutral), youth won or lost money (win trials +$1.00, loss trails -$0.50, total earnings $16.00). We focused on neural response to win or loss (contrasted with neutral) outcomes. Individual contrast images were used to create second-level random effects models using one-sample t-tests for the win > neutral and loss > neutral contrasts. Mean beta weights for the medial PFC (mPFC) and striatal (NAcc, caudate, and putamen) regions of interest (ROIs) were extracted for each contrast. For details and results for each brain regions see Neuropsychopharmacology (2023) 48:623-632; https://doi.org/10.1038/s41386-022-01481-4
Time Frame: Change from pre-treatment (baseline) to post-treatment (12 weeks). Positive values reflect increases in neural response
Population: Participants who completed both baseline and post-treatment fMRI scan (corresponding timepoints for non-anhedonic group). See Neuropsychopharmacology (2023) 48:623-632; https://doi.org/10.1038/s41386-022-01481-4
Measure: Mean (Standard Deviation); unit: Mean beta weights for ROI win > neutral
Arm/Group | Behavioral Activation | Non-anhedonic Adolescent Control Group
Number analyzed (Participants) | 31 | 32
Mean beta weights for ROI win > neutral
  right striatrum | 0.35 (1.41) | -0.31 (1.01)
  left striatum | -0.04 (1.16) | -0.49 (1.59)
  medial pfc | -0.2 (0.9) | -0.17 (1.31)

3. Primary Outcome: Change in Performance (Reward Learning) on the Probabilistic Reward Task (PRT) Computer Task
Description: Each PRT trial begins with a fixation cross (500 ms) followed by a cartoon face without either a mouth or a nose (counterbalanced across subjects and session). After a 500 ms delay, a short or long mouth/nose was presented (100 ms). Participants then indicated whether they saw a short or long mouth or nose. For each block, 40 trials with correct responses resulted in a monetary reward of $0.20. In these cases, participants were presented with a screen that said "Correct! You won 20 cents." While long and short mouths or noses were presented with equal frequency across the block, one length received a reward for correct identification 3x more frequently (i.e., rich stimulus; n=30) than the other (i.e., lean stimulus; n=10). Response bias favoring the rich stimulus was calculated using an established formula (see reference below for details). "Reward Learning" was calculated as the change in response bias score from block 1 to block 2. Higher scores reflect greater reward learning
Time Frame: Change in reward learning from pre-treatment (baseline) to post-treatment (12 weeks).
Population: Participants with usable (passed quality control and not lost due to start of COVID) PRT data at pre- and post-assessment. See Webb et al, Neuropsychopharmacology (2023) 48:623-632; https://doi.org/10.1038/s41386-022-01481-4
Measure: Mean (Standard Deviation); unit: reward learning score
Groups:
- Non-anhedonic Adolescent Control Groupbehavioral Activation: Non-anhedonic (healthy control) adolescents who did not receive behavioral activation
Arm/Group | Behavioral Activation | Non-anhedonic Adolescent Control Groupbehavioral Activation
Number analyzed (Participants) | 32 | 38
reward learning score | 0.08 (0.18) | 0.1 (0.2)

ADVERSE EVENTS:
Time Frame: 12 week behavioral activation trial with 6-month and 1-year follow-up
Arm/Group | Behavioral Activation
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral Activation (N=80)
Suicide attempt (Psychiatric disorders) | 1 (1) — One anhedonic teen attempted suicide (first lifetime attempt) prior to receiving any BA sessions (and was referred to a higher level of psychiatric care after discussions with the study team and participating parents).
Seizure (Nervous system disorders) | 1 (1) — One anhedonic teen in the treatment arm experienced a seizure at home

LIMITATIONS AND CAVEATS:
* Small sample size
* Non-anhedonic adolescents who completed neural and behavioral assessments at timepoints corresponding to the anhedonic group controlled for the effect of repeated assessments and task practice effects. But, a future study with an active control condition is needed to test the specificity of findings to BA vs. other interventions for the treatment of anhedonia in youth
* Generalizability was limited since our sample was largely White and non-Hispanic females

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/25/NCT02498925/Prot_SAP_000.pdf